CLINICAL TRIAL: NCT03173989
Title: Comparison Between Care Strategies for Patients With Osteoarthritis of the Hands Based on the Use of Joint Protection, Assistive Technology and Exercises.
Brief Title: Strategies for Patients With Osteoarthritis, by Using Assistive Technology and Exercises.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Carlos Bandeira de Mello Monteiro, Associate Professor, University of Sao Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 60884416.3.0000.0068
Record Dates: First submitted 2017-05-24; First posted 2017-06-02 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Osteoarthritis Hand
Keywords: osteoarthritis; hand deformities; hand strength; assistive technology; exercise; health education
MeSH Terms: conditions — Osteoarthritis; Hand Deformities; Motor Activity; Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orthosis Exercises Orientation (Experimental): Patients used orthosis, made exercises and received orientation for home.
  Interventions: Device: Orthosis Exercises Orientation
- Orientation (Active Comparator): Patients received orientation for home.
  Interventions: Behavioral: Orientation

INTERVENTIONS:
Device: Orthosis Exercises Orientation — Use of orthosis, exercises and orientation for home.
  Arms: Orthosis Exercises Orientation
Behavioral: Orientation — Orientation for home.
  Arms: Orientation

SUMMARY:
Introduction: Osteoarthritis is a disabling disease that can affect 6% to 12% of the adult population and more than a third of people over 65 years of age. Considering osteoarthritis of hands, existing research about the therapeutic treatment advocates actions such as (1) joint protection, (2) assistive technology and (3) exercises, however, doubts persist as to their effects. Objective: To verify the functional and analgesic effect of joint protection and energy conservation techniques, assistive technology (orthotics and adaptations) and exercises in the treatment of patients with osteoarthritis of the hands. Method: An epidemiological study in which a total sample of patients with knee osteoarthritis will receive joint protection and energy conservation guidelines. Subsequently, the sample will be divided into two groups, group 1 with radiological signs that suggest osteoarthritis of the hands and 2 with patients with radiological signs and symptoms of osteoarthritis of the hands, who present greater functional limitations in the daily life, being eligible for treatment of Rehabilitation, in which will be used orthosis aiming at the relief of pain, stabilization of the affected joints and the prevention of grievance of deformities and orientations of exercises to maintain muscle strength. Participants will be followed up for two years, evaluated with the Disabilities of the Arm, Shoulder and Hand questionnaire (DASH), Stanford Health Assessment Questionnaire (HAQ), palmar grip strength measured with Jamar dynamometer, key pinch strength, three point pinch strength and pulp pinch strength measured with B & L Pinch-gauge dynamometer. The groups will be divided between 1 and 2, the group 1 will be composed of patients who will only perform the orientations informed in the theoretical and practical classes, while the group 2, besides the orientations will receive orthoses with models such as volar hand rest splints, short thumb stabilization splints, and volar finger splints with nocturnal support, aiming at the relief of the pain, stabilization of the affected joints and the prevention of the appearance / aggravation of deformities. Exercise guidelines for maintenance of muscle strength for thumb and fingers will be performed on patients who present significant improvement of pain.

DETAILED DESCRIPTION:
Participants

Were included 200 patients in the group of Bone Metabolic Diseases of the Institute of Orthopedics and Traumatology of the Faculty of Medicine of the University of São Paulo (FMUSP). Were included patients aged between 40 and 80 years, with involvement of osteoarthritis (OA) in the knees and of these, a sample of patients with involvement of the first carpometacarpal, metacarpophalangeal or interphalangeal joint of the thumb and the proximal or distal interphalangeal joint of fingers with from I to III degrees of classification of Kelgreen and Lawrence (KL).

For the calculation of the sample size, a pilot test was performed with 15 subjects and assumed: alpha of 5%, beta of 20% (power = 80%) and difference between the groups of 10% referring to the scores at each scale . With these data, a minimum of 200 individuals was calculated.

Intervention

Participants are patients in an OA treatment program in the Bone Metabolic Diseases group of the Orthopedics and Traumatology Institute of the Faculty of Medicine of the University of São Paulo (FMUSP).

These patients were evaluated for their ability to perform functional activities and anthropometric parameters of upper limbs. The Disability of the Arm, Shoulder and Hand (DASH), the Stanford Health Assessment Questionnaire (HAQ), questionnaires were applied, as well as grip strength measured with Jamar® dynamometer, key pinch, three point pinch, and a pulp pinch measured with B & L Pinch-gauge® dynamometer.

The force was established after arithmetic average of 3 trials. The tests were performed bilaterally. The presence of deformities has also been reported.

The total sample was divided into two groups. Both received guidelines on joint protection and energy conservation, including theoretical and practical classes aimed at protecting all joints that may be affected by OA.

Theoretical classes were carried out through slide presentation with concepts of joint protection, conservation of energy, organization of time, organization of the home and work environment and organization of daily routine. Printed information material was also provided.

The practical classes were carried out in a simulated house, mounted in two rooms of infirmary, suggesting all the environments of a conventional house. Adaptations made by therapists and commercials and conventional objects used in daily living activities were used for the guidelines described above.

The groups were divided between 1 and 2, which was group 1 with patients who presented osteoarthritis in the knees, without specific complaints of hand, but with radiographic findings and group 2 was characterized by patients with radiographic signs and symptoms of hands that presented larger functional limitations in the daily routine or that were eligible for rehabilitation treatment using orthosis models such as resting hand volar splints, thumb stabilization splints or finger volar splints with nocturnal support, aiming at the relief of the pain, stabilization of the affected joints and the prevention of the appearance/aggravation of deformities. Exercise guidelines for maintenance of muscle strength for thumb and fingers were performed in patients who presented significant improvement of pain.

Patients returned for reevaluation at 12 and 24 months after the initial evaluation.

Study Design

Prospective, analytical, experimental, case control study with mixed data collection (prospective and retrospective).

Statistical Analysis

The following variables were considered as dependent variables: HAQ, DASH (general questions, symptons and functions in athletes, performing artists and workers) and dynamometry (manual grip, key pinch, three point pinch and pulp pinch strenght) for the right and left hands. The dependent variables were submitted to ANOVA with factor 2 (Intervention: ortesis, exercises and orientation; orientation) by 8 (group of orientation: 8 different groups of orientation) by 3 (Moment of evaluation: 1- first evaluation [initial], 2- second evaluation [after 1 year], 3- third evaluation [after 2 years]) with repeated measures in the last factor. In order to compare the pain scores in the evaluation moments, the Friedman test was used for the three questions of the DASH's pain module, in a separated moment. Post-hoc comparisons were carried out using Tukey-HSD test (p<0.05).

ELIGIBILITY:
Inclusion Criteria:

* Kellgreen and Lawrence (KL) classification for I to III or painful IV osteoarthritis (with the use of orthoses for analgesia, in this case).
* Capacity to understand and agree to the consent form and questionnaires and evaluations.

Exclusion Criteria:

* Patients who had undergone previous non-medical therapeutic treatment for OA of the hands;
* Who had undergone some surgical procedure in the region or were involved in another clinical trial;
* Patients with rheumatoid arthritis or other rheumatologic disease, any neurological problems.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-08-02 (Actual); Primary Completion 2016-08-05 (Actual); Study Completion 2016-11-05 (Actual)

PRIMARY OUTCOMES:
Patients with orthosis, exercises and orientation will show better results in the evaluation scales regarding strength compared to the group with only orientation. | 2 years
  Strength will be measured dynamometer and compared between groups.

SECONDARY OUTCOMES:
Patients with orthosis, exercises and orientation will show better results in the evaluation scales regarding functionality compared to the group with only orientation. | 2 years
  Functionality will be measured by scales and compared between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos BM Monteiro, Ph.D., Principal Investigator — University of Sao Paulo
Locations (1):
- Escola de Artes,Ciencias e Humanidades da Universidade d Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided